CLINICAL TRIAL: NCT03230448
Title: Study of the Links Between Suicidal Intentionality and Acute Alcoholism
Acronym: ISA
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17-0074; 2017-A00641-52 (Other: ID-RCB)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Suicide, Attempted
Keywords: Acute alcoholism
MeSH Terms: conditions — Suicide, Attempted | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive alcoholism: positive acute alcoholism had questionnaire about suicidal intentionality
  Interventions: Other: questionnaire
- negative alcoholism: negative acute alcoholism had questionnaire about suicidal intentionality
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — after the inclusion patient will answer to a questionnaire about the suicidal intentionality and a second about the alcool consumption

SUMMARY:
There is a strong link between the alcohol consumption and the suicidal risk. Indeed there is an increase of the risk of suicide in case of chronic or acute alcohol consumption. However why the alcohol consumption increase the suicidal risk is unknown.

The hypothesis of this study is that the alcohol consumption induced disinhibition and facilitates the suicide attempt without premeditation

DETAILED DESCRIPTION:
People hospitalized after a suicide attempt will answer to two questionnaires about the suicide intentionality and the acute alcohol consumption.

There is 2 arms:

people doing suicide attempt and with positive level of alcohol (up to 0.1g.L) people doing suicide attempt and with negative level of alcohol

110 patients will be included in this study so 55 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in emergency department for a suicide attempt by voluntary drug intoxication
* speaking and understanding french

Exclusion Criteria:

* Patient who has used other psychoactive substances (attested by toxicological analyzes and / or interrogation)
* Known neurodegenerative pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people hospitalized in the emergency department after a suicide attempt by voluntary drug intoxication
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
compare the score of suicidal intentionality in patient presenting a positive or a negative alcohol level and doing suicide attempt | 15 minutes
  patient will complete the PIERCE questionnaire about the suicidal intentionality

CONTACTS AND LOCATIONS:
Overall Officials: Juliette SALLES, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No